CLINICAL TRIAL: NCT07222072
Title: Methadone to Reduce Chronic Opioid Use After Major Spine Surgery: The MEND Pilot Feasibility Study
Acronym: MEND
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: The MEND Study pilot
Record Dates: First submitted 2025-10-21; First posted 2025-10-29 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Post Operative Pain; Spinal Surgery
Keywords: Methadone; non-opioid; spinal surgery
MeSH Terms: conditions — Pain, Postoperative | interventions — Methadone; Population Groups

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Patients will be randomized 1:1 to postoperative methadone versus placebo on arrival to the operating room. Randomization will occur using a computer-generated randomization system in REDCap, with the sequence of randomly sized blocks pre-determined using the PLAN Procedure in SAS statistical software, stratified by previous history of opioid use (Opioid naïve versus those taking opioids before surgery).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Methadone Group (Active Comparator): Patients randomized to receive post operative methadone
  Interventions: Drug: Methadone
- Patients randomized to receive (blinded) placebo (Placebo Comparator): Patients will receive post operative placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Methadone — Patients randomized to receive (blinded) methadone: 5 mg twice daily on postoperative (post-op) days 1 and 2 followed by 5 mg daily on postop days 3, 4, and 5.
  Other Names: Methadone (Blinded) Group
  Arms: Methadone Group
Drug: Placebo — Patients randomized to receive (blinded) placebo will receive placebo twice daily on day 1 and day 2 and once daily on day 3, 4 and 5. Patients taking preoperative opioids will return to baseline opioid schedule after surgery.
  Other Names: Placebo (Blinded) Group
  Arms: Patients randomized to receive (blinded) placebo

SUMMARY:
The investigators propose a randomized, triple-blinded (patients, investigators, outcomes assessors), placebo-controlled pilot feasibility trial (Methadone to End Narcotic Dependence, MEND trial) to assess the feasibility and safety of postoperative oral methadone in patients undergoing spine surgery and collect preliminary data to inform a larger clinical trial that will test the opioid-sparing effects of methadone at 3 months after spine surgery.

DETAILED DESCRIPTION:
The Centers for Disease Control and Prevention reports a nearly 10-fold increase in the number of deaths from all types of drug overdose over the past 20 years, including 82,000 deaths that occurred in 2022 alone. Prescription opioid medications contribute to drug overdose deaths. In fact, nearly 294,000 people in the US died from a drug overdose involving prescription opioid medications between 1999 and 2022 - a 4-fold increase in prescription drug overdose deaths. Surgery is often the first exposure to opioid medications for many patients. Severe pain after surgery requires potent opioid medications which control pain but includes risk of long-term opioid-dependence. Long-term opioid use and abuse may lead to opioid addiction, overdose and even death.

Patients undergoing spine surgery experience severe postoperative back pain immediately after surgery, which requires treatment with potent opioid medications. Severe pain in the first 1 to 3 days after surgery often develops into chronic back pain, which increases risk for long-term use and abuse of prescription opioid drugs. Importantly, compared with all other surgical procedures, back and spine surgery is associated with the highest risk of long-term use and abuse of prescription opioid medications. Certainly, chronic back pain requires opioid use in approximately 50% of patients at three months after surgery, 40% at six months, 30% at one year, and 17% at two years. A financial burden exists as well. Over the past 10 years, annual prescription opioid expenditures for pain after spine-related surgery increased 660% from $246 million in 1997 to $1.9 billion in 2006. Monthly direct and indirect costs associated with the treatment of postoperative persistent and chronic back pain totaled an average US $3,455 per patient. These data indicate that new approaches that provide effective, long-lasting, and safe treatment of postoperative pain after complex spine surgery while reducing risk of persistent and chronic postoperative pain and prolonged opioid use and reducing cost are needed.

Multiple randomized clinical trials in patients undergoing a variety of surgical procedures have demonstrated that intraoperative methadone significantly reduces postoperative analgesic requirements in the immediate postoperative period, compared to shorter-acting opioids. Methadone is a unique long-acting opioid medication that demonstrates rapid onset and prolonged duration of action with a half-life of 24-36 hours and pain relief lasting 8-12 hours. Like other opioids, methadone activates the mu-opioid receptor, but it also has additional effects on the brain, such as blocking NMDA receptors and reducing reuptake of serotonin and norepinephrine. These actions may help improve recovery by reducing pain sensitivity, preventing tolerance to the medication with euphoric effects, preventing opioid-induced hyperalgesia and opioid tolerance. One investigation studied the impact of methadone on persistent and chronic post-surgical pain in a small randomized controlled trial (RCT) with 66 patients. Participants were randomized to receive either a single intraoperative intravenous dose of methadone (0.2 mg/kg) or intravenous hydromorphone (2 mg). Methadone not only reduced the incidence of post-surgical pain in the study group. but also the percentage of patients who required opioid analgesics at three months (10 versus 41%), suggesting a protective effect against prolonged opioid consumption. Pilot data from another investigation using preoperative oral methadone in patients undergoing cardiac surgery showed reduction in postoperative morphine consumption in the first 24 hours. If acute postoperative pain is reduced, the development of chronic pain may also decrease, as well as the need for long-term opioid therapy, dependence, and abuse.

Although methadone provides effective analgesia for major surgery, a thorough safety assessment of perioperative intravenous methadone is needed. A large retrospective study of 1,478 patients after major spine fusion surgery who received IV methadone (0.13 mg/kg) along with other analgesics, including lidocaine, ketamine, and hydromorphone noted respiratory depression in one-third of patients and hypoxia in nearly 80%. Other concerns include a nearly 60% incidence of electrocardiographic QTc prolongation and 1.1% experienced myocardial infarction (MI) postoperatively. However, there is limited data on the impact of a single perioperative dose of methadone on QTc prolongation. Additional potential complications such as respiratory depression requires further investigation.

If proven safe and effective, postoperative pain therapy with methadone could offer a simple, practical strategy to improve long-term outcomes in this high-risk population undergoing spine surgery. This investigation will the safety and efficacy of postoperative methadone treatment in patients undergoing spine surgery and the opioid-sparing effects of methadone at 3 months after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Adult ≥ 18 years of age
* Scheduled for multilevel lumbar and/or thoracic spine fusion (primary or revision)

Exclusion Criteria:

* <18 or >72 Years of age
* Body Mass Index >40
* Known allergy to methadone
* Pregnant females
* Non-English-speaking patients

Ages: 18 Years to 72 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-11-15 (Actual); Primary Completion 2027-10 (Estimated); Study Completion 2028-10 (Estimated)

PRIMARY OUTCOMES:
Feasibility and Acceptability-Participant Willingness/Recruitment | 7 days
  Willingness of participants to be randomized Indicates acceptability of randomization among eligible patients Outcome Measure: % of eligible patient consenting to randomization
Feasibility and Acceptability-Provider Engagement | 7 days
  Feasibility, acceptability and execution of clinical protocol based on the use of intraoperative IV methadone followed by a postoperative oral methadone regimen following spine surgery will be assessed by yes/no response to the following: Willingness of neurosurgeons/anesthesiologists to buy in to the trial Reflects institutional buy-in and clinical integration potential Outcome Measure: % of surgeons permitting patient enrollment and supporting protocol adherence
Feasibility and Execution-Protocol Compliance and Execution | 7 days
  Feasibility of clinical protocol based on the use of intraoperative IV methadone followed by a postoperative oral methadone regimen following spine surgery will be assessed by yes/no response to the following:
  Compliance with the protocol, including specific study related procedures and timepoints specific to medication administration, adverse event reporting and data collection. Demonstrates deliverability and data reliability Outcome Measure: % adherence to all major protocol steps (drug administration, ECGs, AE reporting, opioid data)
Acceptability and Execution-Baseline Stratification Data | 18 months
  Outcome Measure: % of enrolled patients with prior chronic opioid use
Feasibility and Execution-Follow-Up Completion | 90 days
  Ability to assess primary endpoint (opioid use at 3 months).Measured by response rates to the telephone survey at 3 months

SECONDARY OUTCOMES:
Execution-Collection of Cardiac Rhythm Abnormalities | 18 months
  1) ECG collected on postoperative days 1, 2 and 3. Presence of cardiac arrhythmias (frequent premature ventricular contractions, ventricular arrhythmias) requiring treatment will be collected. An increase in QTc interval >500 ms or >25% from baseline will be compared to baseline ECG,
Execution-Collection of Respiratory Adverse Events | 18 months
  Respiratory depression indicators will be measured every 6 hours.
  1) The presence of any of the following will be considered respiratory depression:
  1. Respiratory rate <8 or oxygen saturation <90% for longer than 5 minutes
  2. Increased oxygen requirement by ≥ 2 L O2 for 15 min
  3. naloxone use. Patients who are receiving
  4. supplemental oxygen
Estimate Reduction in Opioid Use | 90 days
  To estimate reduction in opioid use (Morphine Milligram Equivalents, MME) in the acute postoperative period as a mechanistic indicator for decrease in opioid usage at 3 months.
  Postoperative 5-day opioid requirements assessed by total MME (5 days duration or length of hospitalization, whichever is earlier) will be compared between methadone and placebo groups

OTHER OUTCOMES:
Development of and effective study design | 24 months
  To estimate key design parameters (variability and effect size) of a large clinical trial which will evaluate the reduction in chronic opioid use at 3 months post-surgery. Focusing on estimating parameters that will be needed to appropriately calculate the sample size for a larger trial.

CONTACTS AND LOCATIONS:
Overall Officials: Shobana Rajan, MD, Principal Investigator — The Cleveland Clinic; Andra Duncan, MD, Study Chair — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
The investigator plans to share information by presenting abstract/journal materials pending results.
Supporting Information: Study Protocol, Analytic Code
Time Frame: De-identified data will be available post-analysis in abstract/journal articles.

REFERENCES:
- [Background] Berardino K, Carroll AH, Kaneb A, Civilette MD, Sherman WF, Kaye AD. An Update on Postoperative Opioid Use and Alternative Pain Control Following Spine Surgery. Orthop Rev (Pavia). 2021 Jun 22;13(2):24978. doi: 10.52965/001c.24978. eCollection 2021. PMID 34745473
- [Background] Brummett CM, Waljee JF, Goesling J, Moser S, Lin P, Englesbe MJ, Bohnert ASB, Kheterpal S, Nallamothu BK. New Persistent Opioid Use After Minor and Major Surgical Procedures in US Adults. JAMA Surg. 2017 Jun 21;152(6):e170504. doi: 10.1001/jamasurg.2017.0504. Epub 2017 Jun 21. PMID 28403427
- [Background] Dunn LK, Yerra S, Fang S, Hanak MF, Leibowitz MK, Alpert SB, Tsang S, Durieux ME, Nemergut EC, Naik BI. Safety profile of intraoperative methadone for analgesia after major spine surgery: An observational study of 1,478 patients. J Opioid Manag. 2018 Mar/Apr;14(2):83-87. doi: 10.5055/jom.2018.0435. PMID 29733094
- [Background] Martin BI, Turner JA, Mirza SK, Lee MJ, Comstock BA, Deyo RA. Trends in health care expenditures, utilization, and health status among US adults with spine problems, 1997-2006. Spine (Phila Pa 1976). 2009 Sep 1;34(19):2077-84. doi: 10.1097/BRS.0b013e3181b1fad1. PMID 19675510
- [Background] Luby AO, Alessio-Bilowus D, Hu HM, Brummett CM, Waljee JF, Bicket MC. Trends in Opioid Prescribing and New Persistent Opioid Use After Surgery in the United States. Ann Surg. 2025 Mar 1;281(3):347-352. doi: 10.1097/SLA.0000000000006461. Epub 2024 Aug 1. PMID 39087325
- [Background] Kharasch ED. Intraoperative methadone: rediscovery, reappraisal, and reinvigoration? Anesth Analg. 2011 Jan;112(1):13-6. doi: 10.1213/ANE.0b013e3181fec9a3. No abstract available. PMID 21173206
- [Background] Banks ML, Roma PG, Folk JE, Rice KC, Negus SS. Effects of the delta-opioid agonist SNC80 on the abuse liability of methadone in rhesus monkeys: a behavioral economic analysis. Psychopharmacology (Berl). 2011 Aug;216(3):431-9. doi: 10.1007/s00213-011-2235-2. Epub 2011 Mar 3. PMID 21369752
- [Background] Davidson EM, Coggeshall RE, Carlton SM. Peripheral NMDA and non-NMDA glutamate receptors contribute to nociceptive behaviors in the rat formalin test. Neuroreport. 1997 Mar 3;8(4):941-6. doi: 10.1097/00001756-199703030-00025. PMID 9141069
- [Background] Stubhaug A, Breivik H. Long-term treatment of chronic neuropathic pain with the NMDA (N-methyl-D-aspartate) receptor antagonist ketamine. Acta Anaesthesiol Scand. 1997 Mar;41(3):329-31. doi: 10.1111/j.1399-6576.1997.tb04693.x. No abstract available. PMID 9113174
- [Background] Sotgiu ML, Valente M, Storchi R, Caramenti G, Biella GE. Cooperative N-methyl-D-aspartate (NMDA) receptor antagonism and mu-opioid receptor agonism mediate the methadone inhibition of the spinal neuron pain-related hyperactivity in a rat model of neuropathic pain. Pharmacol Res. 2009 Oct;60(4):284-90. doi: 10.1016/j.phrs.2009.04.002. Epub 2009 Apr 11. PMID 19717013
- [Background] Davis AM, Inturrisi CE. d-Methadone blocks morphine tolerance and N-methyl-D-aspartate-induced hyperalgesia. J Pharmacol Exp Ther. 1999 May;289(2):1048-53. PMID 10215686
- [Background] Mao J, Price DD, Mayer DJ. Mechanisms of hyperalgesia and morphine tolerance: a current view of their possible interactions. Pain. 1995 Sep;62(3):259-274. doi: 10.1016/0304-3959(95)00073-2. PMID 8657426
- [Background] Angst MS, Clark JD. Opioid-induced hyperalgesia: a qualitative systematic review. Anesthesiology. 2006 Mar;104(3):570-87. doi: 10.1097/00000542-200603000-00025. PMID 16508405
- [Background] Kreek MJ, Borg L, Ducat E, Ray B. Pharmacotherapy in the treatment of addiction: methadone. J Addict Dis. 2010 Apr;29(2):200-16. doi: 10.1080/10550881003684798. PMID 20407977
- [Background] Kreutzwiser D, Tawfic QA. Methadone for Pain Management: A Pharmacotherapeutic Review. CNS Drugs. 2020 Aug;34(8):827-839. doi: 10.1007/s40263-020-00743-3. PMID 32564328
- [Background] Gottschalk A, Durieux ME, Nemergut EC. Intraoperative methadone improves postoperative pain control in patients undergoing complex spine surgery. Anesth Analg. 2011 Jan;112(1):218-23. doi: 10.1213/ANE.0b013e3181d8a095. Epub 2010 Apr 24. PMID 20418538
- [Background] Fons RA, Hainsworth KR, Michlig J, Jablonski M, Czarnecki ML, Weisman SJ. Perioperative methadone for posterior spinal fusion in adolescents: Results from a double-blind randomized-controlled trial. Paediatr Anaesth. 2024 May;34(5):438-447. doi: 10.1111/pan.14843. Epub 2024 Jan 30. PMID 38288667
- [Background] Murphy GS, Avram MJ, Greenberg SB, Shear TD, Deshur MA, Dickerson D, Bilimoria S, Benson J, Maher CE, Trenk GJ, Teister KJ, Szokol JW. Postoperative Pain and Analgesic Requirements in the First Year after Intraoperative Methadone for Complex Spine and Cardiac Surgery. Anesthesiology. 2020 Feb;132(2):330-342. doi: 10.1097/ALN.0000000000003025. PMID 31939849
- [Background] Machado FC, Vieira JE, de Orange FA, Ashmawi HA. Intraoperative Methadone Reduces Pain and Opioid Consumption in Acute Postoperative Pain: A Systematic Review and Meta-analysis. Anesth Analg. 2019 Dec;129(6):1723-1732. doi: 10.1213/ANE.0000000000004404. PMID 31743194
- [Background] D'Souza RS, Gurrieri C, Johnson RL, Warner N, Wittwer E. Intraoperative methadone administration and postoperative pain control: a systematic review and meta-analysis. Pain. 2020 Feb;161(2):237-243. doi: 10.1097/j.pain.0000000000001717. PMID 31613867
- [Background] Esfahani K, Tennant W, Tsang S, Naik BI, Dunn LK. Comparison of oral versus intravenous methadone on postoperative pain and opioid use after adult spinal deformity surgery: A retrospective, non-inferiority analysis. PLoS One. 2023 Jul 21;18(7):e0288988. doi: 10.1371/journal.pone.0288988. eCollection 2023. PMID 37478144
- [Background] Eldridge SM, Lancaster GA, Campbell MJ, Thabane L, Hopewell S, Coleman CL, Bond CM. Defining Feasibility and Pilot Studies in Preparation for Randomised Controlled Trials: Development of a Conceptual Framework. PLoS One. 2016 Mar 15;11(3):e0150205. doi: 10.1371/journal.pone.0150205. eCollection 2016. PMID 26978655
- [Background] Moore CG, Carter RE, Nietert PJ, Stewart PW. Recommendations for planning pilot studies in clinical and translational research. Clin Transl Sci. 2011 Oct;4(5):332-7. doi: 10.1111/j.1752-8062.2011.00347.x. PMID 22029804
- [Background] Eldridge SM, Chan CL, Campbell MJ, Bond CM, Hopewell S, Thabane L, Lancaster GA; PAFS consensus group. CONSORT 2010 statement: extension to randomised pilot and feasibility trials. Pilot Feasibility Stud. 2016 Oct 21;2:64. doi: 10.1186/s40814-016-0105-8. eCollection 2016. PMID 27965879
- [Background] Baron RM, Kenny DA. The moderator-mediator variable distinction in social psychological research: conceptual, strategic, and statistical considerations. J Pers Soc Psychol. 1986 Dec;51(6):1173-82. doi: 10.1037//0022-3514.51.6.1173. PMID 3806354
- [Background] Mascha EJ, Dalton JE, Kurz A, Saager L. Statistical grand rounds: understanding the mechanism: mediation analysis in randomized and nonrandomized studies. Anesth Analg. 2013 Oct;117(4):980-994. doi: 10.1213/ANE.0b013e3182a44cb9. Epub 2013 Sep 10. PMID 24023021
- [Background] Austin PC. Balance diagnostics for comparing the distribution of baseline covariates between treatment groups in propensity-score matched samples. Stat Med. 2009 Nov 10;28(25):3083-107. doi: 10.1002/sim.3697. PMID 19757444